CLINICAL TRIAL: NCT05916963
Title: FIRESTONES : Impact of Forced Diuresis on the Residual Fragment Rate After Flexible Ureteroscopy for Destruction of Kidney Stones With Laser: a Randomized Controlled Two-parallel Group Multicenter Trial With Blinding Evaluation
Brief Title: Impact of Forced Diuresis on the Residual Fragment Rate After Flexible Ureteroscopy for Destruction of Kidney Stones With Laser
Acronym: FIREStones
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Tours (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 2022-502890-40-00; DR220258 (Other: Promoter reference)
Record Dates: First submitted 2023-06-14; First posted 2023-06-23 (Actual); Last update posted 2025-11-24 (Actual); Status verified 2025-11

CONDITIONS: Kidney Stone
MeSH Terms: conditions — Kidney Calculi | interventions — Furosemide

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The study will not be blinded except for the outcome assessment: radiologists in charge of interpreting CT-Scans will be blinded.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Furosemide (Experimental): Injection of 40 mg of Furosemide during 10 minutes after the end of the flexible ureteroscopy for destruction of kidney stones with laser.
  Interventions: Drug: Furosemide 40 mg
- Usual care (No Intervention): Usual care, without injection of Furosemide.

INTERVENTIONS:
Drug: Furosemide 40 mg — Injection of 40 mg of Furosemide during 10 minutes after the end of the flexible ureteroscopy for destruction of kidney stones with laser.
  Arms: Furosemide

SUMMARY:
In view of the positive results of the numerous studies conducted on forced diuresis after extra-corporeal lithotripsy, the investigators chose to evaluate forced diuresis by injection of Furosemide associated with intravenous hydration, which has never before been the subject of a specific analysis.

DETAILED DESCRIPTION:
Flexible ureteroscopy is the most common technique to treat kidney stones and is the treatment of choice in France.

Kidney stones destruction requires its laser pulverization into small fragments in order to remove them through the ureter or improve their spontaneous expulsion along the urinary tract. However, most of the time, all the micro-fragments and dust created during stone destruction cannot be extracted using our surgical tools, and may stay intra-renally at the end of the procedure. Although these micro-fragments are expected to disappear spontaneously by the natural flushing and peristalsis of the upper urinary tract, they remain at risk of stagnation that could be the nest of new aggregation and stone formation.

Adjuvant treatments (such as forced diuresis, inversion or mechanical pressure) were previously described to improve the expulsion of stone fragments after extra-corporeal shock wave lithotripsy.

Nevertheless, the impact of adjuvant treatment after flexible ureteroscopy remains unclear and mainly theoretical.

In view of the positive results of the numerous studies conducted on forced diuresis after extra-corporeal lithotripsy, the investigators chose to evaluate forced diuresis by injection of Furosemide associated with intravenous hydration, which has never before been the subject of a specific analysis.

Loop diuretics (including Furosemide) significantly increase diuresis, which results in a greater flow of urine into the renal cavities, improving the chances of evacuating the residual fragments of the stone destroyed during flexible ureteroscopy, before they can sediment in the fundus of the renal calices or in the pyelon. Therefore, the investigators hypothesize that a forced diuresis with an injection of Furosemide at the end of ureteroscopy could improve the micro-fragments and stones dust clearance.

ELIGIBILITY:
Inclusion Criteria:

* Patients ≥ 18 years old and < 80 years old
* With the need to perform a flexible ureteroscopy with destruction of the kidney stones with laser
* Participants covered by or entitled to social security
* Written informed consent obtained from the participant
* Ability for participant to comply with the requirements of the study

Exclusion Criteria:

* Persons covered by articles L1121-5 to L1121-8 of the CSP (corresponding to all protected persons: pregnant women, parturients, nursing mothers, persons deprived of their liberty by judicial or administrative decision, minors, and persons subject to a legal protection measure: guardianship or trusteeship)
* Contra-indication to Furosemide:

  * Hyper-sensitivity to the active substance or one of the excipients
  * Hyper-sensitivity to Sulfonamide
  * Renal failure with oligo-anuria refractory to Furosemide
  * Hypokalemia < 3,5 mmol/L
  * Severe hyponatremia
  * Hypovolemia with or without hypotension or dehydration
  * Ongoing hepatitis, hepatic insufficiency severe and hepatic encephalopathy
* Patient having Furosemide as usual treatment
* Patient requiring an injection of Aminoside or Vancomycin before or during the procedure
* Participation in other interventional research with an investigational drug or medical device

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 374 (Estimated)
Dates: Start 2024-01-04 (Actual); Primary Completion 2026-04-03 (Estimated); Study Completion 2026-04-03 (Estimated)

PRIMARY OUTCOMES:
Rate of stone free patients | At 3 months
  Rate of stone-free patients 3 months after a flexible ureteroscopy for renal stone laser destruction, evaluated on the low dose abdomino-pelvic CT-Scan.
  A centralized review of the images will be performed by two specialized radiologists, in a blind and crossed way to allow a homogenization of the results

SECONDARY OUTCOMES:
Rate of urinary infection | From baseline to 30 days
  Rate of post-operative urinary tract infection will be assessed within 30 days after surgery on the combination of:
  * Fever higher than 38.5°C and/or,
  * Chills and/or,
  * Clinical symptoms (supra-pubic pain, dysuria, pollakiuria, urgency, urinary burning, back pain radiating to the genitals, hematuria) and/or
  * Positive urine culture with a significant bacteriuria threshold defined as bacteriuria ≥10^5 UFC/mL with one or two bacterial species.
Pain in a scale | During the hospital stay
  Post-operative pain will be assessed on numerical pain scale in the recovery room, in the service and at the discharge. Pain scale is from 0 (no pain) to 10 (as bad as it could be nothing else matters)
Opioid consumption | During the hospital stay, an average of 1 day
  The use of opioids will be reported
Number of participants with adverse events | From baseline to 3 months, an average of 1 day
  Number of participants with Furosemide adverse events

CONTACTS AND LOCATIONS:
Locations (9):
- France (9):
  - CHU d'Angers, Angers
  - Hospices Civils de Lyon, Lyon
  - CHU de Nice, Nice
  - CHU de Nîmes, Nîmes
  - CHU de Rennes, Rennes
  - CHU de Rouen, Rouen
  - CHU de Toulouse, Toulouse
  - Clinique La Croix du Sud, Toulouse
  - CHRU de Tours, Tours

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Letouche ML, Giraudeau B, Agier MS, Bruyere F. FIRE Stones: impact of forced diuresis on the residual fragment rate after flexible ureteroscopy for destruction of kidney stones with laser-protocol for a randomized controlled two-parallel group multicenter trial with blinding evaluation. Trials. 2024 Jul 4;25(1):455. doi: 10.1186/s13063-024-08309-0. PMID 38965611